CLINICAL TRIAL: NCT03179891
Title: A Multicenter, Open Label, Crossover Study to Assess the Pharmacokinetics and Safety of Diazepam Buccal Soluble Film (DBSF) in Adult Subjects With Epilepsy
Brief Title: Study of Diazepam Buccal Film Administered in the Interictal and in the Ictal-Periictal States to Adults With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Collaborators: inVentiv Health Clinical (Other); Covance (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 160326
Record Dates: First submitted 2017-05-26; First posted 2017-06-07 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Epilepsy
Keywords: Interictal; Ictal/peri-ictal
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: This was a multicenter, open-label study comprised of 2 treatment periods with a minimum 14 days washout between the 2 treatment periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interictal Period (Experimental): All subjects received 12.5 mg DBF during the interictal state.
  Interventions: Drug: Diazepam Buccal Film 12.5 mg
- Ictal/Peri-ictal Period (Experimental): All subjects received 12.5 mg DBF during the ictal/peri-ictal state.
  Interventions: Drug: Diazepam Buccal Film 12.5 mg

INTERVENTIONS:
Drug: Diazepam Buccal Film 12.5 mg — All subjects received a single dose of DBF 12.5 mg during the interictal state and during the ictal/peri-ictal state with at least 14 days washout between the 2 treatment periods
  Other Names: DBF 12.5mg

SUMMARY:
This Phase 2 open-label, two-way study was conducted in adult subjects with epilepsy who were on stable regimens of anti-epileptic drugs (AEDs) and who were admitted to an Epilepsy Monitoring Unit (EMU), General Clinical Research Center (GCRC), or similar facility for evaluation of their seizures. All subjects received a single DBF 12.5 mg dose during the Interictal State and a single DBF 12.5 mg dose during the Ictal/peri-ictal state with at least 14 days washout between the 2 doses.

DETAILED DESCRIPTION:
This was a Phase 2 multicenter, open-label, two-way study conducted in adult subjects to assess the bioavailability, pharmacokinetics, and safety of DBF during the Interictal Period and during the Ictal/peri-ictal Period, with a minimum of 14 days of washout between periods. Subjects had a clinical diagnosis of epilepsy (with generalized tonic-clonic seizures or focal seizures with impaired awareness) who were on stable regimens of anti-epileptic drugs and were scheduled for admission to an EMU, GCRC, or similar facility for evaluation.

All subjects were to receive a single 12.5-mg dose of study drug, without regard to meals, during both Interictal Period and Ictal/peri-ictal Period. The treatment was identical for both periods. Treatment sequence was not randomized. The interictal period and ictal/peri-ictal could occur in either order as determined by seizure occurrence.

Interictal Period: Subjects were considered to be in an interictal state if an interval of at least 3 hours had elapsed since any clinically observable postictal signs or symptoms (from the last observed seizure) and the subject had been seizure-free over this period. Subjects on electroencephalogram (EEG) video monitoring were to be considered to be in an interictal state if an interval of at least 3 hours had elapsed since there were any postictal electrical findings on EEG.

Ictal/peri-ictal Period: For the purposes of this study, the ictal state was defined as an ongoing clinically observable seizure or seizure activity as verified via EEG. The periictal state was defined clinically as the subject's immediate postictal state following a generalized tonic-clonic (GTC) seizure or focal seizure with impaired awareness, and within 5 minutes following the last clonic jerk. For subjects on EEG video monitoring, the periictal state was to be defined as less than 5 minutes after cessation of seizure activity as verified via EEG.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects meeting all of the following criteria may be included in the study:

1. Subjects scheduled for admission to the institution's EMU, GCRC (General Clinical Research Center) or similar facility for evaluation within 28 days.
2. Male and female subjects between 18 to 65 years of age, inclusive.
3. Subjects having a body weight of ≥ 40 kg to 111 kg.
4. Subjects have a clinical diagnosis of epilepsy and are scheduled to be admitted to an Epilepsy Monitoring Unit (EMU) for extracranial video-Electroencephalogram (EEG) recording of a seizure event for evaluation of their epilepsy.
5. Subjects have an average frequency of > 1 seizure every 3 days or > 10 seizures / month as documented by seizure diaries dispensed at the Screening Visit and verified prior to initiation of Period A or Period B.
6. Female subjects have a negative serum pregnancy test at Screening. Female subjects of childbearing potential (i.e., not surgically sterile or 2 years postmenopausal) must have a negative pregnancy test at screening and a partner who is sterile, agree to abstinence, be practicing double barrier contraception or using an FDA approved contraceptive (e.g., licensed hormonal or barrier methods) for greater than 2 months prior to screening visit and commit to an acceptable form of birth control for the duration of the study and for 30 days after participation in the study.
7. Subjects are currently receiving at least one antiepileptic medication.
8. Subjects or subject's legally authorized representative (LAR) must be willing and able to complete informed consent/assent and HIPAA authorization.
9. Subjects must agree and must be willing to comply with all required study procedures while in the EMU or GCRC.
10. Ability to comprehend and be informed of the nature of the study, as assessed by the PI or Sub-Investigator.
11. Ability to consume standard meals.
12. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded:

1. Subjects having a progressive neurological disorder such as brain tumor, demyelinating disease, or degenerative central nervous system (CNS) disease that is likely to progress in the next 12 months.
2. Subjects having respiratory failure (or is at risk for respiratory failure) or other severe cardiorespiratory disease with New York Heart Association Class III or IV functional status, or requires supplemental oxygen.
3. Female subjects who are lactating or positive serum pregnancy test (ß-hCG) at screening for female subjects ≥12 years of age.
4. Subjects with severe psychiatric disease that in the Investigator's judgment would prevent the patient's successful completion of the study.
5. Subjects who have an episode of status epilepticus, as determined by the Principal Investigator/Sub-Investigator, at any time during Period B (EMU, GCRC or similar facility Visit
6. Subjects with known history or presence of any clinically significant hepatic (e.g. hepatic impairment), renal/genitourinary (renal impairment, kidney stones), psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the Principal Investigator/Sub-Investigator and confirmed by Sponsor via written communication prior to subject enrollment.
7. Subjects with any clinically significant illness other than epilepsy within 30 days prior to first dosing, as determined by the Principal Investigator/Sub-Investigator.
8. Subjects with any significant physical or organ abnormality as determined by the Principal Investigator/Sub-Investigator.
9. Subjects with any significant lesion of the oral cavity or having oral prophylactic procedures within 30 days prior to first dosing.
10. Subjects with a QTc interval QTcF>450 msec for males and QTcF>470 msec for females on screening ECG, unless determined as not clinically significant by the Investigator.
11. Subjects with a positive test result for any of the following: drugs of abuse (amphetamines, cocaine, opiates, or phencyclidine), a positive breath alcohol test.
12. Subjects with a known history or presence of: a. Alcohol abuse or dependence within one year prior to first drug administration; b. Drug abuse or dependence; c. Hypersensitivity or idiosyncratic reaction to diazepam, its excipients, sodium phosphates; and/or related substances, e.g. benzodiazepines; d. Glaucoma (open or acute narrow angle); e. Severe allergic reactions (e.g. anaphylactic reactions, angioedema
13. Subjects who have participated in another clinical trial or who received an investigational drug within 30 days prior to first drug administration or 5 half-lives of the investigational drug-whichever is the longer period.
14. Blood or plasma donation within 30 days prior to Screening
15. Subjects not willing or unable to tolerate blood draws.
16. Subjects who have received any other dosage form of diazepam or benzodiazepines within 2 weeks prior to entering Period A or Period B.
17. Consumption of alcohol within 48 hours before dosing and food or beverages containing grapefruit, star fruit, Seville oranges, and/or pomelo or their derived products (e.g., fruit juice) within 10 days prior to first drug administration.
18. Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g. cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, or HIV antivirals) and strong inducers of CYP enzymes (e.g. glucocorticoids, St. John´s Wort, or rifampicin) in the previous 30 days before first drug administration [barbiturates, carbamazepine, and phenytoin are allowed since these are common AEDs (Anti-epileptic drugs)].
19. Use of any monoamine oxidase (MAO) inhibitors (e.g. phenelzine, tranylcypromine), phenothiazines (chlorpromazine) within 30 days prior to first drug administration.
20. Employee or immediate relative of an employee of the investigator, MonoSol Rx LLC, any of its affiliates or partners, or inVentiv Health.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Slatko, Study Director — Aquestive Therapeutics
Locations (11):
- United States (11):
  - Arizona Health Sciences Center, Tucson, Arizona
  - Rancho Research Institute, Downey, California
  - Yale University School of Medicine-Comprehensive Epilepsy Center, New Haven, Connecticut
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Onsite Clinical Solutions LLC, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Austin Epilepsy Care Center, Austin, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned enrollment was 40 adult male and female subjects with a clinical diagnosis of epilepsy requiring admission to an epilepsy monitoring unit, a general clinical research center, or similar facility for evaluation of seizures. A minimum of 30 subjects was expected to complete the study.
Pre-assignment Details: A total of 35 subjects were enrolled to receive a 12.5-mg dose of study drug during both the interictal and the ictal/peri-ictal period which occurred in either order as determined by seizure occurrence.
Groups:
- Interictal State First, Then Ictal/Peri-ictal State: Subjects received DBF 12.5 mg during the Interical State first and then during the Ictal/Peri-ictal State with at least 14 days washout between the 2 periods.
- Ictal/Peri-Ictal State First, Then Interictal State: Subjects received DBF 12.5 mg during the ictal/peri-ictal state first and then during the interictal state with at least 14 days washout between the 2 periods.
Period: First Intervention
Arm/Group | Interictal State First, Then Ictal/Peri-ictal State | Ictal/Peri-Ictal State First, Then Interictal State
Started | 13 | 22
Completed | 11 | 20
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Unspecified reason | 1 | 0
Not completed — Protocol Violation | 0 | 1
Period: Second Intervention (After 14 Days)
Arm/Group | Interictal State First, Then Ictal/Peri-ictal State | Ictal/Peri-Ictal State First, Then Interictal State
Started | 11 | 20
Completed | 11 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Thirty-five subjects were enrolled to receive DBF 12.5 mg in both Interictal and Peri-ictal period with order determined by seizure occurrence. Four subjects withdrew after receiving their first dose; 2 subjects in the Interictal Period and 2 subjects in the Ictal/peri-ictal period.
Groups:
- Adult Subjects With Epilepsy: Adult subjects with epilepsy admitted to an Epilepsy Monitoring Unit to receive a single 12.5 mg DBF dose during the Ictal Phase and during the Interictal/Peri-ictal Phase with at least 14 days between the 2 periods
Arm/Group | Adult Subjects With Epilepsy
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants] — Population: Thirty-five adult subjects with epilepsy received at least 1 dose of study drug and were included in the analysis of safety.
  participants
    United States | 35
Height [Mean (Standard Deviation); unit: cm] | 165.64 (10.81)
Weight [Mean (Standard Deviation); unit: kg] | 79.24 (19.58)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.84 (7.01)

OUTCOME MEASURES:

1. Primary Outcome: Tmax Pharmacokinetic EndPoints
Description: Observed time to reach maximum drug concentration (Tmax)
Time Frame: -2 to 0, 0.25, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 192, 240 hours
Population: The pharmacokinetic analysis set comprised only those subjects who contributed a valid pharmacokinetic profile for the given analysis and whose predose concentration of the relevant analyte did not exceed 5% of the subsequent Cmax.
Measure: Median (Full Range); unit: hours
Groups:
- Interictal State: Single 12.5-mg dose of Diazepam Buccal Film administered during the interictal state
  Adult subjects with epilepsy
- Ictal/Peri-ictal State: Single 12.5-mg dose of Diazepam Buccal Film administered during the ictal/peri-ictal state
  Adult subjects with epilepsy
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 32 | 24
hours | 1.000 [0.249 to 4.017] | 0.525 [0.250 to 2.033]

2. Primary Outcome: Cmax Pharmacokinetic EndPoints
Description: Observed Peak Drug Concentration (Cmax)
Time Frame: -2 to 0, 0.25, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 192, 240 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Interictal State: Single 12.5 mg dose of Diazepam Buccal Film administered during the interictal state
  Adult subjects with epilepsy
- Ictal/Peri-ictal State: Single 12.5 mg dose of Diazepam Buccal Film administered during the ictal/peri-ictal state.
  Adult subjects with epilepsy
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 32 | 24
ng/mL | 230.32 (89.00) | 209.49 (120.18)

3. Primary Outcome: Area Under the Plasma Concentration Curve Pharmacokinetic EndPoints
Description: Area under the Plasma Concentration -time curve from time zero until the last measured time (AUC0-t)
Time Frame: -2 to 0, 0.25, 0.5, 1, 2, 4, 8, 24, 48, 96, 144, 192, 240 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 32 | 24
h*ng/mL | 560.18 (219.70) | 498.78 (319.09)

4. Secondary Outcome: Usability Endpoint - Successful Insertion/Placement of the Diazepam Buccal Film (DBF) on First Attempt
Description: Number of subjects with unsuccessful insertion/placement of the DBF on first attempt at administration Number of subjects with successful insertion/placement of the DBF on first attempt at administration
  Placement is judged to be successful when film adheres to the center of buccal mucosa of either right or left cheek.
  Unsuccessful placements were followed by a subsequent successful insertion/placement of DBF
Time Frame: Subject was observed for 15 minutes after initial film placement/adhesion
Population: Safety Population comprising all subjects who received at least 1 dose of study drug (Diazepam Buccal Film).
Measure: Count of Participants; unit: Participants
Groups:
- Interictal State: Single 12.5-mg dose of Diazepam Buccal Film administered during the interictal state.
  Adult subjects with epilepsy
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 33 | 33
Participants
  Unsuccessful insertion/placement | 0 | 2
  Successful insertion/placement | 33 | 31

5. Secondary Outcome: Usability Endpoint: Swallowing the Film Before Complete Disintegration/Dissolution
Description: Was the film noted to have been swallowed by the subject ? Yes No
  Subjects were instructed to swallow any remnants of film still present in oral cavity 15 minutes after initial film placement.
  Results include subjects who swallowed film at any point during the 15 minutes immediately after initial film placement.
Time Frame: Subject was observed for 15 minutes immediately following DBF placement/adhesion
Population: Safety Population comprising all subjects who received at least 1 dose of study drug (Diazepam Buccal Film).
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 33 | 33
Participants
  Yes-DBF was Swallowed | 4 | 2
  No-DBF was not Swallowed | 29 | 31

6. Secondary Outcome: Usability Endpoint: Retention of Diazepam Buccal Film (DBF) From Placement to Complete Disintegration
Description: Was the DBF spit out or blown out by the subject after placement on buccal mucosa or did the subject chew, talk, or move the DBF prior to complete disintegration/dissolution? Yes No
Time Frame: Subject was observed for 15 minutes immediately following DBF placement/adhesion
Population: Safety Population comprising all subjects who received at least 1 dose of study drug (Diazepam Buccal Film).
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 33 | 33
Participants
  Yes-DBF was spit out/blown out | 0 | 3
  No-DBF was not spit out/blown out | 33 | 30

7. Secondary Outcome: Usability Endpoint: Exit of Saliva During the Time the Diazepam Buccal Film (DBF) Was Adhered to Buccal Mucosa
Description: The observer documented if any saliva was seen to exit the mouth during the time the DBF was adhered to buccal mucosa
Time Frame: Subject was observed for 15 minutes immediately following DBF placement/adhesion
Population: Safety Population comprising all subjects who received at least 1 dose of study drug (Diazepam Buccal Film).
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 33 | 33
Participants
  Yes, saliva exited the mouth | 0 | 2
  No, saliva did not exit mouth | 33 | 31

8. Secondary Outcome: Usability Endpoint: Amount of Saliva That Exited the Mouth After Film Placement
Description: If Yes - saliva exited the mouth during the time, estimate in milliliters of the amount of saliva that exited the mouth after DBF placement on the buccal surface
Time Frame: Subject was observed for 15 minutes immediately following DBF placement/adhesion
Population: Safety Population comprising all subjects who received at least 1 dose of study drug (Diazepam Buccal Film).
Measure: Count of Participants; unit: Participants
Arm/Group | Interictal State | Ictal/Peri-ictal State
Number analyzed (Participants) | 33 | 33
Participants
  Participants with 0 mL saliva exiting the mouth | 33 | 31
  Participants with 1 mL saliva exiting the mouth | 0 | 1
  Participants with 2 mL saliva exiting the mouth | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study for each subject (approximately 1 month for each subject - beginning with the first DBF dose until 14 ± 2 days following the second DBF dose).
Groups:
- Interictal State (Period A): Single 12.5-mg dose of Diazepam Buccal Film administered during the interictal state.
  Adult subjects with epilepsy
- Ictal/Peri-ictal State (Period B): Single 12.5-mg dose of Diazepam Buccal Film administered during the ictal/peri-ictal state.
  Adult subjects with epilepsy
Arm/Group | Interictal State (Period A) | Ictal/Peri-ictal State (Period B)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 12/33 | 14/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interictal State (Period A) (N=33) | Ictal/Peri-ictal State (Period B) (N=33)
HOSPITALIZATION DUE TO SEIZURE CLUSTER (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interictal State (Period A) (N=33) | Ictal/Peri-ictal State (Period B) (N=33)
Complex Partial Seizures (Nervous system disorders) | 9 (9) | 14 (14)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Generalized tonic-clonic seizure (Nervous system disorders) | 1 (6) | 1 (3)
Seizure (Nervous system disorders) | 1 (2) | 1 (4)
Somnolence (Nervous system disorders) | 2 (3) | 0 (0)
Seizure cluster (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results were included as confidential information and required written sponsor approval.

DOCUMENTS (2):
  • Study Protocol (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03179891/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03179891/SAP_001.pdf